CLINICAL TRIAL: NCT05038579
Title: Clinical Validation of a Cognitive Stimulation Platform for Individuals With Dementia - Musiquence
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidade da Madeira (Other)
Collaborators: Instituto São João de Deus (Unknown); Casa de Saúde Câmara Pestana (Unknown); Centro Social e Paroquial da Ribeira Brava (Unknown); Associação de Desenvolvimento Comunitário do Funchal, Centro de Dia Lugar de Memórias (Unknown)
Responsible Party: Principal Investigator, Sergi Bermúdez i Badia, Associate Professor at the University of Madeira and Senior Researcher at NOVA-LINCS, Universidade da Madeira
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 9/CEUMA/2021
Record Dates: First submitted 2021-05-04; First posted 2021-09-09 (Actual); Last update posted 2021-09-09 (Actual); Status verified 2021-09

CONDITIONS: Dementia
Keywords: Dementia; Cognitive stimulation; Musiquence; Music; Reminiscence; Augmented Reality
MeSH Terms: conditions — Dementia

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Musiquence (Experimental): Dementia group was involved in a 14-session customized cognitive stimulation program, using Musiquence.
  Interventions: Procedure: Musiquence

INTERVENTIONS:
Procedure: Musiquence — The participants performed a customized cognitive stimulation program, that was implemented in an augmented reality format, using Musiquence.

SUMMARY:
Dementia is a neurodegenerative syndrome that leads to cognitive deficits and, consequently, affects functionality and quality of life.

This study will explore the clinical impact of a customized cognitive stimulation program, using Musiquence.

DETAILED DESCRIPTION:
Dementia is a clinical syndrome characterized by a progressive and irreversible deterioration of cognitive functioning that impairs behavioral and functional domains. Within non-pharmacological approaches, Cognitive Stimulation Therapy (CST) is the most studied and well-established intervention for individuals with mild to moderate dementia. The underlying assumptions behind cognitive-based interventions of CST are:

1. IwD can benefit from cognitive stimulation if mobilized relatively preserved cognitive functions (e.g., crystallized abilities such as semantic memory and verbal skills), and;
2. Even in advanced age, exposure to enriched environments (i.e., socially and cognitively challenging) can enhance cognitive reserve and neuroplasticity.

Concerning the first assumption of cognitive-based interventions (a1), it is known that even in moderate to advanced stages of dementia, musical memory is one of the abilities that remain intact. It is hypothesized that music processing abilities precede the development of lexical language functions. This hypothesis is corroborated by findings that demonstrate that IwD are still responsive to music even when unable to communicate verbally or recognize words. Additionally, music is frequently associated with life experiences. Also, literature has reported that memories associated with specific music would be recollected longer than memories with no association to music; this suggests that using music as a reminiscence element on cognitive stimulation programs can have a promising effect on cognition. According to the second assumption of CST (a2), facilitating an enriching environment for IwD using, for , music and reminiscence elements could impact cognitive reserve and neuroplasticity.

In this context, Ferreira et al. developed a platform - Musiquence - that incorporates music and reminiscence in cognitive stimulation activities for IwD. Musiquence allows the gamification and personalization of 6 types of activities:

* Reality Orientation - a quiz-like activity that includes date and time information.
* Creative Drawings - a puzzle-like game in which the participant draws the missing pieces.
* Activities of Daily Living (ADL) - a puzzle-like game in which the participants have to perform a set of chores (i.e., brush the teeth), and the missing pieces are completed with real physical objects (i.e., toothpaste).
* Search Objects activity - exploration game in which the participants must find hidden images (e.g., cats) that are only visible through a virtual magnifying glass.
* Knowledge Quiz - participants must select the correct answer to a question among incorrect ones.
* Association activity - participants must categorize the items according to the instructions. For example, separate cars from motorcycles and locate them in the correct container.

The platform is compatible with different technologies that allow adaptation to the patients' needs (motor difficulties, vision problems, tremble). Cognitive stimulation content can be personalized to the user since the caregivers can add text, images, and music when creating the tasks.

ELIGIBILITY:
Inclusion Criteria:

* Mild to moderate stage of dementia (with formal diagnosis);
* Ability to move upper limbs;
* Maintained auditory acuity;
* Relatively preserved language skills.

Exclusion Criteria:

* Moderate to severe depressive symptomatology;
* Moderate to severe anxious symptomatology;
* Bedridden.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2019-09-01 (Actual); Primary Completion 2020-11-30 (Actual); Study Completion 2021-02-28 (Actual)

PRIMARY OUTCOMES:
Mini-Mental State Examination (Cognitive Screening) (MMSE) | Baseline, Post-intervention (7 weeks), Follow-up (3 months)
  Change from baseline in the MMSE. Minimum of 0 points and maximum of 30 points. Higher scores mean better outcomes.
Alzheimer's Disease Assessment Scale - Cognitive Scale (ADAS - Cog) | Baseline, Post-intervention (7 weeks), Follow-up (3 months)
  Change from baseline in the ADAS-Cog. Minimum of 0 points and maximum of 68 points. Higher scores mean worse outcomes.

SECONDARY OUTCOMES:
Quality of Life - Alzheimer's Disease (QoL - AD) | Baseline, Post-intervention (7 weeks), Follow-up (3 months)
  Change from baseline in the QoL - AD. Minimum of 0 points and maximum of 52 points. Higher scores mean better outcomes.
Kettler Laurent Thierreau (KLT) | Baseline, Post-intervention (7 weeks), Follow-up (3 months)
  Change from baseline in the KLT. Minimum of 0 points and maximum of 100 ponints.Higher scores mean worse outcomes.
Symbol Search - Weschler Adult Inteligence Scale 3rd edition (SR) | Baseline, Post-intervention (7 weeks), Follow-up (3 months)
  Change from baseline in the SR Minimum of 0 points and maximum of 10 points.. Higher scores mean better outcomes.
Digital Symbol Coding - Weschler Adult Inteligence Scale 3rd edition (DSC) | Baseline, Post-intervention (7 weeks), Follow-up (3 months)
  Change from baseline in the DSC. Minimum of 0 points and maximum of 10 points. Higher scores mean better outcomes.
Semantic and Phonemic Verbal Fluency (SPVF) | Baseline, Post-intervention (7 weeks), Follow-up (3 months)
  Change from baseline in the SPVF. Minimum of 0 points and no maximum. Higher scores mean better outcomes.
Adults and Older Adults Functional Assessment Inventory (IAFAI) | Baseline, Post-intervention (7 weeks), Follow-up (3 months)
  Change from baseline in the IAFAI. Minimum of 0 points and maximum of 100 points. Higher scores mean worse outcomes.
Cornell Scale for Depression in Dementia | Baseline, Post-intervention (7 weeks), Follow-up (3 months)
  Change from baseline in the Cornell Scale for Depression in Dementia. Minimum of 0 points and maximum of 38 points. Higher scores mean worse outcomes.
Rating Anxiety in Dementia (RAID) scale. | Baseline, Post-intervention (7 weeks), Follow-up (3 months)
  Change from baseline in the RAID. Minimum of 0 points and maximum of 54 points. Higher scores mean worse outcomes.

CONTACTS AND LOCATIONS:
Locations (1):
- Universidade da Madeira, Funchal, Madeira, Portugal

DOCUMENTS (1):
  • Study Protocol (2021-05-27): https://cdn.clinicaltrials.gov/large-docs/79/NCT05038579/Prot_000.pdf